CLINICAL TRIAL: NCT05734157
Title: Chansu Vascular Technologies Everolimus-Coated Balloon Percutaneous Transluminal Angioplasty Catheter First-in-Human Clinical Investigation
Brief Title: CVT-SFA First in Human Trial for Treatment of Superficial Femoral Artery or Proximal Popliteal Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP1109
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Femoral Artery Stenosis; Popliteal Artery Stenosis; Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: TP1109; CVT-SFA; Femoral Artery Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Everolimus-coated balloon (Experimental): Treatment of patients with de-novo or post-PTA occluded/stenotic or re-occluded/restenotic lesions in femoropopliteal arteries with a drug-coated balloon.
  Interventions: Device: Peripheral PTA with a drug coated balloon

INTERVENTIONS:
Device: Peripheral PTA with a drug coated balloon — Peripheral artery angioplasty

SUMMARY:
The CVT-SFA Trial investigates the inhibition of restenosis using the CVT Everolimus-coated PTA Catheter in the treatment of de-novo occluded/ stenotic or re-occluded/restenotic superficial femoral or popliteal arteries.

DETAILED DESCRIPTION:
The CVT-SFA Trial is a prospective, multi-center, open, single arm study enrolling subjects with de-novo or post-PTA occluded/stenotic or re-occluded/ restenotic lesions (excluding in-stent lesions) ≤150mm in length in femoropopliteal arteries with reference vessel diameters of 4-6mm, receiving up to two (2) CVT Everolimus-coated PTA Catheters to establish blood flow and to maintain vessel patency.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or his/her legally authorized representative provides written informed consent prior to any clinical investigation related procedure, as approved by the appropriate Ethics Committee of the respective clinical site.
3. Subject must agree to undergo all clinical investigation plan-required follow-up visits and examinations.
4. Subjects with symptomatic leg ischemia, requiring treatment of SFA or popliteal (P1 segment) artery.
5. De novo or restenotic lesion(s) >70% within the SFA and popliteal arteries in a single limb which are ≥3 cm and ≤15 cm in cumulative total length (by visual estimation). Lesion must be at least 2 cm from any stented area.
6. Subject is willing to comply with the required follow up visits, testing schedule and medication regimen.
7. Successful wire crossing of lesion.
8. Target vessel reference diameter ≥4 mm and ≤6 mm (by visual estimation).
9. Target lesion(s) can be treated with a maximum of two (2) CVT Everolimus-coated PTA Catheters.
10. At least one patent (less than 50% stenosis) tibio-peroneal run-off vessel confirmed by baseline angiography or prior MR angiography or CT angiography.
11. Life expectancy >1 year
12. Rutherford classification of 2, 3 or 4.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Co-existing clinically significant aneurismal disease of the abdominal aorta, iliac or popliteal arteries.
3. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
4. Known intolerance to study medications, everolimus or contrast agents.
5. Doubts in the willingness or capability of the subject to allow follow-up examinations.
6. Subject is actively participating in another investigational device or drug study.
7. History of hemorrhagic stroke within 3 months of procedure.
8. Previous or planned surgical or interventional procedure within 30 days of index procedure.
9. Prior vascular surgery of the target lesion.
10. Lesion length is <3 cm or >15 cm or there is no normal proximal arterial segment in which duplex ultrasound velocity ratios can be measured.
11. Known inadequate distal outflow.
12. Significant inflow disease.
13. Acute or sub-acute thrombus in target vessel.
14. Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloons, brachytherapy, lithotripsy).
15. Outflow arteries (distal popliteal, anterior or posterior tibial or peroneal arteries) with significant lesions (≥ 50% stenosis) may not be treated during the same procedure.
16. Treatment of the contralateral limb during the same procedure or within 30 days of the study procedure.
17. Rutherford classification of 0, 1, 5 or 6
18. Presence of prohibitive calcification that precludes adequate PTA treatment.
19. Subjects held in custody in an institution by official or court order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- France (4):
  - Polyclinique Les Fleurs, Ollioules
  - Hôpital Paris Saint Joseph, Paris
  - Hôpital Nord Laennec - CHU de Nantes, Saint-Herblain
  - Clinique Pasteur, Toulouse
- Germany (4):
  - Institut für Radiologie, Kinderradiologie und interventionelle Therapie, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - DIAKO Krankenhaus Flensburg, Flensburg
  - Romed Klinikum Rosenheim, Rosenheim

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total seventy-five (75) subjects were enrolled in the CVT-SFA study at eight (8) investigational sites in Europe between February 17, 2022, and September 01, 2022.
Groups:
- Everolimus-coated Balloon: The Chansu Vascular Technologies (CVT) Everolimus-coated PTA Catheter is an angioplasty catheter designed to facilitate percutaneous treatment of subjects with documented symptomatic occlusion and/or >70% stenosis of the SFA or popliteal (P1 segment) artery.
  The CVT Everolimus-coated PTA Catheter is comprised of two main components:
  1. A CE-marked, commercially-available PTA balloon catheter designed to treat peripheral vascular artery lesions. The PTA catheters are also previously cleared by FDA for peripheral (PTA) angioplasty indications.
  2. A drug coating comprised of an approved, commercially-available active pharmaceutical agent (API) mixed with an approved commercially-available excipi Theent. active pharmaceutical agent is the drug everolimus, in crystalline form, and it is applied onto the balloon using a glycerol ester excipient. Everolimus, like sirolimus, is an mTOR inhibitor drug with cytostatic properties. Everolimus is currently used in CE mark and FDA approved coronary drug-eluting stents [Promus (Boston Scientific), Xience (Abbott Vascular), Synergy (Boston Scientific)].
Period: Overall Study
Arm/Group | Everolimus-coated Balloon
Started | 75
Completed | 66
Not Completed | 9
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Telephone call | 3

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 62
  More than one race | 0
  Unknown or Not Reported | 13
Hypertension [Count of Participants; unit: Participants] | 58

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Freedom of Major Adverse Event (MAE) Rate
Description: Composite rate of cardiovascular death, index limb amputation and ischemia-driven target lesion revascularization (TLR).
Time Frame: 6 months post procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 72

2. Primary Outcome: The Primary Effectiveness Endpoint: Patency (Freedom From Restenosis, Freedom From Ischemia-driven TLR)
Description: Freedom from restenosis as determined by duplex ultrasonography (DUS) (peak systolic velocity ratio (PSVR) ≤2.4 or ≤50% stenosis) and freedom from ischemia-driven target lesion revascularization (TLR).
Time Frame: 6 months post procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 68
Participants | 63

3. Secondary Outcome: Rate of Major Adverse Event (MAE)
Description: Composite rate of cardiovascular death, index limb amputation and ischemia-driven Target Lesion Revascularization (TLR). The time frame for "In hospital" refers to time from procedure to discharge. This timeframe is different for every enrolled subject. The subject is discharged at the treating physician's discretion based on their specific treatment needs.
Time Frame: In Hospital
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 0

4. Secondary Outcome: Rate of Major Adverse Event (MAE)
Description: Composite rate of cardiovascular death, index limb amputation and ischemia-driven Target Lesion Revascularization (TLR).
Time Frame: 30 Days Post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 1

5. Secondary Outcome: Rate of Major Adverse Event (MAE)
Description: Composite rate of cardiovascular death, index limb amputation and ischemia-driven Target Lesion Revascularization (TLR).
Time Frame: 12 months Post-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 72
Participants | 67

6. Secondary Outcome: Rate of Occurrence of Arterial Thrombosis of the Treated Segment
Description: Rate of occurrence arterial thrombosis of the treated segment as determined by QVA
Time Frame: 12months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 0

7. Secondary Outcome: Rate of Ipsilateral Embolic Events of the Study Limb
Description: This end point was to asses the Rate of Ipsilateral Embolic Events of the Study Limb.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 2

8. Secondary Outcome: Rate of Clinically-driven Revascularization
Description: This end point was to asses the Rate of Clinically-driven Revascularization.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 74
Participants | 2

9. Secondary Outcome: Rate of Clinically-driven Revascularization
Description: This end point was to asses the Rate of Clinically-driven Revascularization.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 72
Participants | 4

10. Secondary Outcome: Patency Rate
Description: The patency results achieved in the CVT-SFA Study translate into meaningful patient benefits as demonstrated by the improvement of secondary outcomes measures.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 67
Participants | 61

11. Secondary Outcome: Rate of Vascular Access Site Complication
Description: Rate of vascular access site complication defined as the combined rate of hematoma, AV fistula or a pseudoaneurysm that required intervention, such as surgical repair or transfusion, prolonged hospital stay, or required a new hospital admission.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 2

12. Secondary Outcome: Lesion Success
Description: Lesion success (per device), defined as achievement of a final in-lesion residual diameter stenosis of <50% (by QA), using any device after wire passage through the lesion. Pre- and post-dilatation of the lesion with a non-study device is considered part of assigned device treatment.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 86
Lesions | 85

13. Secondary Outcome: Technical Success
Description: Technical success (per device), defined as achievement of a final in-lesion residual diameter stenosis of <50% (by QA), using the CVT Everolimus-coated PTA Catheter without a device malfunction after wire passage through the lesion. Pre- and postdilatation are considered part of assigned device treatment.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Number analyzed (lesions) | 86
lesions | 85

14. Secondary Outcome: Clinical Success
Description: Clinical success (per subject) defined as technical success without the occurrence of major adverse events (MAE) during the procedure.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 75

15. Secondary Outcome: Procedural Success
Description: Procedural success (per subject) defined as lesion success without the occurrence of major adverse events during procedure.
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants | 75

16. Secondary Outcome: Change in Ankle-Brachial Index (ABI)
Description: Change in Ankle-Brachial Index (ABI) is calculated as the difference between the ABI values at baseline and at follow-up visits. ABI is measured using a Doppler ultrasound or Oscillo metric method to assess peripheral arterial function. A change of ≥0.1 in ABI values from baseline to follow-up is considered clinically significant. The data presented in the Outcome Measure table reflects the percentage of participants who experienced a significant change in ABI from baseline.
Time Frame: Discharge
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 71
Participants | 61

17. Secondary Outcome: Change in Ankle-Brachial Index (ABI)
Description: as for outcome 16
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 71
Participants | 69

18. Secondary Outcome: Change in Ankle-Brachial Index (ABI)
Description: as for outcome 16
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 71
Participants | 61

19. Secondary Outcome: Walking Impairment Questionnaire - Patient Perceived Change in Walking Difficulty
Description: The WIQ (Walking Impairment Questionnaire) score is a numerical representation of a person's walking capacity, derived from their responses to a series of questions about walking difficulty. Individuals are asked to rate degree of difficulty of various activities with responses ranging from 0 (lowest possible function) to 4 (highest possible function). Questions within each category are based on degree of difficulty, according to approximate number of feet, stairs, or miles per hour for distance, stair-climbing, and speed scores, respectively. Scores are then divided by maximum number of points and presented on a scale of 0% to 100%, where 0% represents lowest possible score (i.e., answering "unable" for all questions in that category) and 100% represents the highest possible score (i.e., indicating "none" with regard to difficulty for all questions in that category). A higher score indicates less difficulty with walking, while a lower score signifies greater difficulty with walking.
Time Frame: Pre-Procedure to 6 months and 12 months
Population: Number of participants who completed the Patient Reported Outcome (PRO) tool at each study time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
score on a scale
  Pre procedure | 31.3 (29.7)
  6 months: number analyzed (Participants) | 72
  6 months | 78.0 (36.9)
  12 months: number analyzed (Participants) | 67
  12 months | 80.8 (35.6)

20. Secondary Outcome: Walking Impairment Questionnaire - Patient Perceived Change in Walking Speed
Description: The WIQ (Walking Impairment Questionnaire) score is a numerical representation of a person's walking capacity, derived from their responses to a series of questions about walking difficulty. Individuals are asked to rate the degree of difficulty of various activities with responses ranging from 0 (lowest possible function) to 4 (highest possible function). Questions within each category are based on the degree of difficulty, according to the approximate number of feet, stairs, or miles per hour for the distance, stair-climbing, and speed scores, respectively. Scores are then divided by the maximum number of points and presented on a scale of 0% to 100%, where 0%represents the lowest possible score (i.e., answering "unable" for all questions in that category) and 100% represents the highest possible score (i.e., indicating "none" with regard to difficulty for all questions in that category). Higher scores signify less difficulty in maintaining speed while walking.
Time Frame: Pre-Procedure to 6 months and 12 months
Population: Number of participants who completed the Patient Reported Outcome (PRO) tool at each study time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
score on a scale
  Pre procedure | 19.0 (16.7)
  6 months: number analyzed (Participants) | 72
  6 months | 46.6 (31.5)
  12 months: number analyzed (Participants) | 67
  12 months | 44.9 (31.7)

21. Secondary Outcome: Walking Impairment Questionnaire - Patient Perceived Change in Walking Impairment
Description: The WIQ (Walking Impairment Questionnaire) score is a numerical representation of a person's walking capacity, derived from their responses to a series of questions about walking difficulty. Individuals are asked to rate the degree of difficulty of various activities with responses ranging from 0 (lowest possible function) to 4 (highest possible function). Questions within each category are based on the degree of difficulty, according to the approximate number of feet, stairs, or miles per hour for the distance, stair-climbing, and speed scores, respectively. Scores are then divided by the maximum number of points and presented on a scale of 0% to 100%, where 0%represents the lowest possible score (i.e., answering "unable" for all questions in that category) and 100% represents the highest possible score (i.e., indicating "none" with regard to difficulty for all questions in that category). A higher score indicates less perceived walking impairment.
Time Frame: Pre-Procedure to 6 months and 12 months
Population: Number of participants who completed the Patient Reported Outcome (PRO) tool at each study time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
score on a scale
  Pre procedure | 75.9 (17.6)
  6 months: number analyzed (Participants) | 72
  6 months | 85.3 (17.8)
  12 months: number analyzed (Participants) | 67
  12 months | 89.9 (12.9)

22. Secondary Outcome: Walking Test: Change in Walking Distance
Description: The Walking Test is a standard test used to evaluate functionality in patients with peripheral artery disease (PAD). This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline to 6 months and 12 months
Population: Number of participants who completed the Patient Reported Outcome (PRO) tool at each study time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 73
meters
  Baseline: number analyzed (Participants) | 25
  Baseline | 231.3 (93.6)
  6 months: number analyzed (Participants) | 22
  6 months | 382.8 (151.7)
  12 months: number analyzed (Participants) | 26
  12 months | 399.6 (138.6)

23. Secondary Outcome: Treadmill Test: Change in Walking Distance
Description: Treadmill walking test is a standard test used to evaluate functionality in patients with peripheral artery disease (PAD).
Time Frame: Baseline to 6 months and 12 months
Population: Number of participants who completed the Patient Reported Outcome (PRO) tool at each study time point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
meters
  Baseline: number analyzed (Participants) | 42
  Baseline | 80.9 (52.8)
  6 months: number analyzed (Participants) | 37
  6 months | 104.0 (72.7)
  12 months: number analyzed (Participants) | 34
  12 months | 106.0 (74.6)

24. Secondary Outcome: Change in Rutherford Classification
Description: Participants were graded using the Rutherford Classification, which stages PAD based on symptoms and clinical findings.
  Class 0 asymptomatic , normal treadmill or reactive hyperemia test. Class 1 mild claudication completes treadmill exercise; AP after exercise > 50 mm Hg but at least 20 mm Hg lower than resting value.
  Class 2-3 more severe symptoms cannot complete standard treadmill exercise, and AP after exercise < 50 mm Hg.
  Class 4 critical limb ischemia resting AP < 40 mm Hg, flat or barely pulsatile ankle or metatarsal PVR; TP < 30 mm Hg.
  Class 5 minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia and resting AP < 60 mm Hg, ankle or metatarsal PVR flat or barely pulsatile; TP < 40 mm Hg. The lower the RB Class the better the outcome.
Time Frame: Pre-procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 75
Participants
  Class 0 | 0
  Class 1 | 0
  Class 2 | 12
  Class 3 | 53
  Class 4 | 9
  Class 5 | 1
  Class 6 | 0
  Not Done | 0

25. Secondary Outcome: Change in Rutherford Classification
Description: as for outcome 24
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 74
Participants
  Class 0 | 51
  Class 1 | 6
  Class 2 | 7
  Class 3 | 6
  Class 4 | 0
  Class 5 | 0
  Class 6 | 0
  Not Done | 4

26. Secondary Outcome: Change in Rutherford Classification
Description: as for outcome 24
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus-coated Balloon
Number analyzed (Participants) | 72
Participants
  Class 0 | 51
  Class 1 | 3
  Class 2 | 5
  Class 3 | 7
  Class 4 | 0
  Class 5 | 0
  Class 6 | 0
  Not Done | 6

ADVERSE EVENTS:
Time Frame: Baseline to 12 months
Arm/Group | Everolimus-coated Balloon
All-Cause Mortality (participants affected / at risk) | 3/75
Serious Adverse Events (participants affected / at risk) | 37/75
Other Adverse Events (participants affected / at risk) | 51/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus-coated Balloon (N=75)
Anemia (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 7
Death during heart surgery (Cardiac disorders) | 1
Heart attack (Cardiac disorders) | 1
Partial Infarct (Cardiac disorders) | 1
Right ventricular implant repair (Cardiac disorders) | 1
Colon tumor (Gastrointestinal disorders) | 1
Epigastric pain (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Inflammatory bladder (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cancer (General disorders) | 1
Terminal cancer (General disorders) | 2
Aneurysm spurium (Injury, poisoning and procedural complications) | 2
Distal embolism (Injury, poisoning and procedural complications) | 1
Revascularization (Injury, poisoning and procedural complications) | 5
Spinal contusions (Musculoskeletal and connective tissue disorders) | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Parkinson's Disease (Nervous system disorders) | 1
Stenosis, non-study limb (General disorders) | 15
Stenosis, non-study vessel (General disorders) | 1
Stenosis, non-target lesion (General disorders) | 2
Stenosis, target vessel (General disorders) | 1
Cystitis (Renal and urinary disorders) | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1
Lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal resection (squamous cell cancer) (Skin and subcutaneous tissue disorders) | 1
Glaucoma surgery (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus-coated Balloon (N=75)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
CRP increase at discharge (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 3
Irregular heartrate (Cardiac disorders) | 1
Thoracic pain (Cardiac disorders) | 1
Burning pain in esophagus (Gastrointestinal disorders) | 1
Esophageal reflux (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Allergy to medication (General disorders) | 2
Angiography performed (General disorders) | 5
Bruises easily (General disorders) | 1
Bruising/hemotoma over body (General disorders) | 1
Calf claudication (General disorders) | 1
Calf pain (General disorders) | 3
Deep vein thrombosis, non-study limb (General disorders) | 1
Diabetes mellitus II (General disorders) | 1
Distal arteriopathy (General disorders) | 1
Dizzyness (General disorders) | 1
Glaucoma (General disorders) | 1
Groin bleeding (General disorders) | 1
Groin/scrotum hematoma (non-study limb) (General disorders) | 1
Haematoma, right arm (General disorders) | 1
Haematoma, wrist (General disorders) | 1
Hip pain (General disorders) | 2
Knee injury (General disorders) | 1
Knee pain (General disorders) | 4
Leg claudication, non-study limb (General disorders) | 1
Leg oedema, both legs (General disorders) | 1
Leg pain (General disorders) | 3
Lower body/limbs hot (General disorders) | 1
Lower leg swelling (General disorders) | 1
Necrosectomy, heel (General disorders) | 1
Oedema, non-study limb (General disorders) | 1
Pain, non-study limb (General disorders) | 1
Polyneuropathy, non-study limb (General disorders) | 1
Stenosis, non-TL (General disorders) | 5
Stenosis, non-study limb (General disorders) | 2
Swollen knee (General disorders) | 1
TL occlusion, no action taken (General disorders) | 5
Teeth extraction (General disorders) | 1
Tension headache (General disorders) | 1
Tingling/numbing foot (General disorders) | 1
Toe pain (General disorders) | 1
Vertigo (General disorders) | 1
Covid (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
AV fistula post-dilatation (Injury, poisoning and procedural complications) | 1
Bleeding at groin puncture site (Injury, poisoning and procedural complications) | 1
Distal embolism (Injury, poisoning and procedural complications) | 1
Groin pain (Injury, poisoning and procedural complications) | 2
Groin pain at puncture site (Injury, poisoning and procedural complications) | 2
Hematoma at puncture site (Injury, poisoning and procedural complications) | 2
Pain in lower leg (Injury, poisoning and procedural complications) | 1
Perforation from guidewire (Injury, poisoning and procedural complications) | 1
Superficial thrombosis (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Disc prolapse (Musculoskeletal and connective tissue disorders) | 1
Sciatica pain (Musculoskeletal and connective tissue disorders) | 1
Spinal canal stenosis (Musculoskeletal and connective tissue disorders) | 1
Chronic kidney insufficiency (Renal and urinary disorders) | 1
Skin tumor (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT05734157/Prot_SAP_000.pdf